CLINICAL TRIAL: NCT03875287
Title: A Phase I Dose-Escalation Study of E7727, an Oral Cytidine Deaminase Inhibitor (CDAi) With Oral Decitabine in Subjects With Solid Tumors
Brief Title: Dose-Escalation Study of E7727, an Oral Cytidine Deaminase Inhibitor With Oral Decitabine in Subjects With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry); Stand Up To Cancer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: J18115; IRB00182038 (Other: JHM IRB); ASTX727 (Other: Astex Pharmaceuticals)
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Decitabine; cedazuridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Decitabine and Cedazuridine (Experimental): Treatment will be administered on an outpatient basis. Cycle length is 28 days. The dose of cedazuridine is fixed at 100mg and the dose and duration of decitabine will vary depending on when a patient enters the study.
  Interventions: Drug: Decitabine; Drug: Cedazuridine

INTERVENTIONS:
Drug: Decitabine — DOSING REGIMEN(S):
  Level -1 10mg daily days 1-4
  Level 1 10mg daily days 1-5
  Level 2 15mg daily days 1-5
  Level 3 20mg daily days 1-5
  Level 4 25 mg daily days 1-5
  Other Names: Dacogen
Drug: Cedazuridine — DOSING REGIMEN(S):
  Level -1 100mg daily days 1-4
  Level 1 100mg daily days 1-5
  Level 2 100mg daily days 1-5
  Level 3 100mg daily days 1-5
  Level 4 100mg daily days 1-5

SUMMARY:
This is a phase 1 study of the combination of cedazuridine with decitabine in patients with solid tumors. At least 6 patients will be enrolled per treatment level to assess optimal hypomethylation and toxicity (up to 35 patients total).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have advanced, unresectable, and/or metastatic solid tumor malignancy that is histologically or cytologically confirmed.
* Patients must have received at least 2 lines of therapy in the advanced/metastatic setting (if 2 lines exist) and have no other possible therapies or refuse therapies that have shown clinical benefit for their condition.
* ECOG performance status <1
* Ability to understand and the willingness to sign a written informed consent document.
* Patients must have measurable disease
* Ability to swallow oral medications

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 3 weeks
* Participants may not be receiving any other investigational agents.
* Active hepatitis B or hepatitis C infection.
* Active or untreated gastric or duodenal ulcer
* Symptomatic bowel obstruction within 3 months prior to screening visit.
* Symptomatic ascites in the last 4 weeks

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of combination cedazuridine with decitabine as assessed by number of participants who experience adverse events | up to 2 years
  Number of participants who have experienced grade 3 or higher adverse events, as defined by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0)
Maximum Tolerated Dose (MTD) as determined by number of participants with of dose limiting toxicities (DLT) | up to 2 years
  Maximum tolerated dose will be determined by the maximum dose at which the least number of participants experience dose-limiting toxicity. The dose limiting toxicity is defined using the Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Pharmacokinetics of ASTX727 in solid tumor patients as measured by total exposure | Day 2
  Total exposure will be calculated as area under the plasma concentration-time curve (AUC) by using non-compartmental methods (Winonlin, version 5.3 or newer) and/or compartmental modeling (Adapt II, release 4.0)
Pharmacokinetics of ASTX727 in solid tumor patients as measured by maximum concentration (Cmax) | Day 2
  Cmax (mmol/L) is defined as the maximum concentration of ASTX727 in blood.
Pharmacokinetics of ASTX727 in solid tumor patients as measured by time to maximum concentration (Tmax) | Day 2
  Tmax (minutes) is defined as the time to reach maximum concentration of ASTX727 in blood.
Objective response rate (ORR) in solid tumor patients who are treated with ASTX727 | up to 2 years
  Proportion of participants who had measurable disease at baseline and have been re-evaluated after at least 1 cycle of therapy with observed reduction in tumor burden as defined by RECIST 1.1: Complete response (CR)= disappearance of all target lesions, Partial response (PR)= at least 30% decrease in sum of diameters of target lesions

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland